CLINICAL TRIAL: NCT01633632
Title: Hatha Yoga as an Adjunct to Cognitive Behavioral Therapy for Smoking Cessation
Brief Title: Hatha Yoga for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-16438/13-16721
Record Dates: First submitted 2012-07-02; First posted 2012-07-04 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Yoga; Cognitive behavioral therapy
MeSH Terms: conditions — Smoking Cessation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cognitive behavioral therapy (Active Comparator): This group will receive a standardized, 8-session cognitive behavioral therapy course that is offered to the public at our practice.
  Interventions: Behavioral: Cognitive behavioral therapy
- Cognitive behavioral therapy + yoga (Experimental): This group will receive the standardized, 8-session cognitive behavioral therapy course + 8 sessions of Hatha yoga.
  Interventions: Behavioral: Hatha yoga; Behavioral: Cognitive behavioral therapy
- Hatha yoga (Experimental): This group will receive 8 sessions of Hatha yoga and printed materials to assist with their quit attempt
  Interventions: Behavioral: Hatha yoga

INTERVENTIONS:
Behavioral: Hatha yoga — 30 minutes of instruction in Hatha yoga will be provided for 8 sessions.
  Arms: Cognitive behavioral therapy + yoga; Hatha yoga
Behavioral: Cognitive behavioral therapy — 8-sessions of cognitive behavioral therapy will be provided following a standardized curriculum.
  Arms: Cognitive behavioral therapy; Cognitive behavioral therapy + yoga

SUMMARY:
The purpose of this study is to determine whether Hatha Yoga can improve the chances of a successful smoking quit attempt.

DETAILED DESCRIPTION:
While many smoking cessation interventions have been studied, even the most successful interventions result in less than 40% abstinence from smoking at 6 months. Most people attempt to quit multiple times before maintaining long-term abstinence from tobacco. Research into interventions to improve quit rates and decrease smoking prevalence is a high priority for multiple organizations. Yoga is an attractive non-pharmacological option because it can be used safely during pregnancy and lactation, can be combined with other pharmacologic and non-pharmacologic treatments, and can be continued well past the smoking cessation date to combat withdrawal symptoms and cravings. There is a critical need for innovative and effective methods for tobacco control that focus on both prevention and cessation.

This project will be broken into two stages. The first stage will aim to pilot test yoga techniques for feasibility and acceptability. Recruitment and retention strategies will be tested and participant satisfaction will be evaluated. Preliminary measures of smoking abstinence and withdrawal symptoms will be conducted.

The second stage of this study will be a randomized trial to compare smoking abstinence with cognitive behavioral therapy (CBT), CBT + yoga, or yoga alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Smoker of 5 or more cigarettes per day
* Willing and physically able to participate in yoga
* Not currently practicing Hatha yoga.

Exclusion Criteria:

* Use of smokeless tobacco

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Point prevalence abstinence from smoking | End of intervention (week 7)
  Abstinence from smoking as measured by expired carbon monoxide at the end of the 7-week intervention.

SECONDARY OUTCOMES:
Abstinence from smoking | 3 and 6 months
  Prolonged abstinence defined as no smoking after the identified "quit date" and point prevalence abstinence (no smoking in the past 7 days) will be measured. Measured by self-report.
Change in weight | End of intervention (week 7)
  Change in weight from baseline to week 7
Signs and symptoms of nicotine withdrawal | Weeks 1-7 during intervention period
  Survey will be administered weekly during class sessions

CONTACTS AND LOCATIONS:
Overall Officials: Amy Mayer, OTD, OTR/L, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Result] Burns TL, Mayer AE, Washington-Krauth SM, Walters RW, Arouni AJ. Design and Feasibility of a Hatha Yoga Intervention for Smoking Cessation. Journal of Smoking Cessation 2014; doi:10.1017/jsc.2014.21.